CLINICAL TRIAL: NCT05383872
Title: A Pivotal Study to Evaluate the Safety and Effectiveness of Exablate Model 4000 Using Microbubble Resonators to Temporarily Mediate Blood-Brain Barrier Disruption (BBBD) for Liquid Biopsy in Subjects With GlioBlastoma Brain Tumors
Brief Title: Blood-Brain Barrier Disruption (BBBD) for Liquid Biopsy in Subjects With GlioBlastoma Brain Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BT015
Record Dates: First submitted 2022-04-25; First posted 2022-05-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Glioma; Liquid Biopsy
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Exablate BBBD (Experimental): Using Exablate Model 4000 Type 2 for liquid biopsy in subjects with Glioblastoma
  Interventions: Device: Focused Ultrasound (Exablate Model 4000)

INTERVENTIONS:
Device: Focused Ultrasound (Exablate Model 4000) — BBB opening via Exablate Type 2 system with microbubble resonators and drawing blood before and after opening

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of targeted blood brain barrier disruption with Exablate Model 4000 Type 2.0/2.1 for liquid biopsy in subjects with suspected Glioblastoma brain tumors

DETAILED DESCRIPTION:
This is a prospective, multi-center, pivotal clinical trial to evaluate the safety and efficacy of targeted blood brain barrier disruption using Exablate Model 4000 Type 2 for liquid biopsy in subjects with suspected Glioblastoma brain tumors. The study will be conducted at up to 25 centers in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects18-80 years of age who are able and willing to give informed consent, or whose legally authorized representative is willing to consent on their behalf
2. Subjects with stereotactically-targetable suspected new or recurrent glioblastoma tumor on pre-operative brain imaging scans
3. Subjects that are scheduled, or will be scheduled within 4 weeks, for surgical resection or biopsy per standard clinical tumor care
4. Karnofsky Performance Score >70
5. Able to communicate sensations during the Exablate BBBD procedure

Exclusion Criteria:

1. Subjects with inoperable tumors (e.g., tumor originating from the deep midline, thalamus, midbrain, cerebellum or brainstem)
2. Multifocal tumors
3. Tumor morphology or other imaging findings that precludes the ability to sonicate the tumor volume (including significant tumor volume outside the treatment envelope or tumor volume that exceeds the maximum sonication volume allowed, i.e. currently 110 ccs at the treatment volume level). Concern for adequate tumor coverage by sonication based on tumor morphology should be discussed with the Sponsor.
4. MRI or clinical findings of:

   1. Active or chronic infection(s) or inflammatory processes
   2. Acute or chronic hemorrhages, specifically any lobar microbleeds, and no siderosis, amyloid angiopathy, or macro-hemorrhages
   3. Intracranial thrombosis, vascular malformation, cerebral aneurysm or vasculitis
5. MR non-compatible metallic implants in the skull or the brain or the presence of unknown MR unsafe devices
6. Significant cardiac disease or unstable hemodynamic status

   1. Documented myocardial infarction within six months of enrollment
   2. Unstable angina on medication
   3. Unstable or worsening congestive heart failure
   4. Documented left ventricular ejection fraction below the lower limit of normal
   5. History of a hemodynamically unstable cardiac arrhythmia
   6. Cardiac pacemaker
7. Uncontrolled hypertension (systolic > 180 and diastolic BP > 120 on medication)
8. Undergoing anti-coagulant or anti-platelet therapy, or using medications known to increase risk of hemorrhage within washout period prior to treatment (i.e., antiplatelet or vitamin K inhibitor anticoagulants within 7 days, non-vitamin K inhibitor anticoagulants within 72 hours, or heparin-derived compounds within 48 hours of treatment).
9. History of bleeding disorder, coagulopathy or a history of spontaneous hemorrhage or evidence of increased risk of bleeding
10. Abnormal coagulation profile (Platelets < 80,000, PT >14, PTT >36, or INR > 1.3)
11. Known cerebral or systemic vasculopathy
12. Significant depression and at potential risk of suicide
13. Known sensitivity/allergy to gadolinium or DEFINITY/DEFINITY RT,
14. Active seizures despite medication treatment (defined as >1 seizure per week) which could be worsened by disruption of the blood brain barrier
15. Active drug or alcohol disorder which have a higher risk for seizures, infection and/or poor executive functioning
16. Known positive HIV status, which can lead to increased entry of HIV into the brain parenchyma leading to HIV encephalitis
17. Potential blood-borne infections which can lead to increased entry to brain parenchyma leading to meningitis or brain abscess
18. Any contraindications to MRI scanning, including:

    1. Large subjects not fitting comfortably into the scanner
    2. Difficulty lying supine and still for up to 3 hours in the MRI unit or claustrophobia
19. Impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
20. Severe Respiratory Illness: chronic pulmonary disorders (e.g., severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area), subjects with a history of severe drug allergies, severe asthma or hay fever, or multiple allergies where the benefit/risk of administering DEFINITY/DEFINITY RT is considered unfavorable by the study physicians in relation to the product labeling for DEFINITY/DEFINITY RT
21. Currently in a clinical trial involving an investigational product or non-approved use of a drug or device
22. Pregnancy or Lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Through study completion, up to 1 year
  All adverse events and/or Serious Adverse Events will be documented and reported according to CTCAE
Correlation with Tumor Tissue | Up to 3 hours Post-BBBD
  To demonstrate there is a correlation between patterns obtained in the panel of biomarkers evaluated in the resected tumor tissue and/or biopsy and blood sample collected post-BBBD

SECONDARY OUTCOMES:
Circulating Free DNA | Up to 3 hours Post-BBBD
  To demonstrate that there is at least a 2-fold increase in circulating free DNA following blood brain barrier disruption (BBBD)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (16):
  - University of California, Los Angeles, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California San Francisco, San Francisco, California
  - UF Health Shands Hospital, Gainesville, Florida
  - Miami Cancer Institute at Baptist Health, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Maryland, Baltimore & The University of Maryland Medical System, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - NYU Grossman School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Texas, Southwestern, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - West Virginia University Rockefeller Neuroscience Center, Morgantown, West Virginia
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No